CLINICAL TRIAL: NCT06266676
Title: The Effects of Heart Surgery Nursing Mobile Micro-course in Perioperative Registered Nurse.
Brief Title: Mobile Micro-course Impact on Perioperative RNs in Heart Surgery Nursing.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ting-Fang Yeh (Other)
Responsible Party: Sponsor-Investigator, Ting-Fang Yeh, Registered Nurse, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202301775B1
Record Dates: First submitted 2024-01-13; First posted 2024-02-20 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: periOperative; Cardiac Surgical Procedures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- micro-course (Experimental): The experimental group adopts micro-course instruction, providing self-directed learning through online asynchronous courses, with instructional content delivered through short videos created by the researcher.
  Interventions: Other: micro-course
- slide presentation (Active Comparator): The control group, on the other hand, employs a unidirectional teaching method by the instructor, offering self-directed learning through online asynchronous courses, primarily using researcher-created online presentations.
  Interventions: Other: slide presentation

INTERVENTIONS:
Other: micro-course — The experimental group adopts micro-course instruction, providing self-directed learning through online asynchronous courses, with instructional content delivered through short videos created by the researcher.
  Arms: micro-course
Other: slide presentation — Provide online presentations.
  Arms: slide presentation

SUMMARY:
The goal of this clinical trialis to compare in learning effectiveness of nurses. The main questions it aims to answer are:

1. Can the "Micro-course" teaching enhance the awareness of cardiac surgery nursing among operating room nurses?
2. Can the "Micro-course" teaching boost the learning motivation and engagement of operating room nurses?
3. What is the satisfaction level of nurses regarding the use of "Micro-course" in cardiac surgery nursing?
4. What are the relevant factors influencing the effectiveness of the "Micro-course" teaching intervention?

Participants will be divided into two groups. The control group will receive online presentations, while the experimental group will engage in mobile learning combined with micro-courses. Both groups of participants will undergo instruction through asynchronous online courses.

ELIGIBILITY:
Inclusion Criteria:

1. Currently engaged in clinical surgical nursing and possess a valid nursing license.
2. Individuals who have not received training for cardiac surgery scrub nursing or who have received such training but have not worked as a cardiac surgery scrub nurse for more than two years.
3. Nurses involved in the collaborative use of personnel during operating room duty.

Exclusion Criteria:

1. Nursing supervisors at the level of charge nurse or higher.
2. Nurses exclusively engaged in local anesthesia surgical nursing.
3. Nurses primarily engaged in waiting room, recovery room, and anesthesia nursing.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Cognitive scale | Before the experiment commenced, all participants underwent a uniform pre-test. A post-test was administered one week after the conclusion of the course. A second post-test was conducted four weeks after the course concluded (this served as a delayed ass
  The cognitive scale was self-designed by the author after referencing textbooks and journal articles. It is divided into four dimensions based on teaching topics, with a total of 15 single-choice questions to assess nurses' cognition of cardiac surgery. Each correct answer earns 1 point, with higher scores indicating higher levels of cognition.
motivation scale | Before the experiment started, all participants underwent a standardized pre-test. A post-test was conducted one week after the conclusion of the course
  The scale consists of 12 items and employs a four-point Likert scale for scoring, ranging from 4 points for "strongly agree" to 1 point for "strongly disagree." Higher scores indicate stronger learning motivation.
Engagement Scale | One week after the course concluded, measurements were taken.
  This scale comprises a total of 10 items, scored using a four-point Likert scale, ranging from 4 points for "strongly agree" to 1 point for "strongly disagree." Higher scores indicate a higher level of learning engagement among the research subjects.

SECONDARY OUTCOMES:
learning satisfaction | One week after the course concluded, measurements were taken.
  There are a total of 10 questions, along with 2 open-ended questions. Scoring for this scale is based on a four-point Likert scale, ranging from 4 points for "strongly agree" to 1 point for "strongly disagree." Higher scores indicate higher levels of satisfaction with learning among nurses.

CONTACTS AND LOCATIONS:
Locations (1):
- ChangGungMH, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No